CLINICAL TRIAL: NCT06177808
Title: Assessment of Cutting-Balloon Angioplasty With Novel Bioabsorbable Polymer-Coated, Everolimus-Eluting Stent in the Treatment of Calcified Coronary Lesions Guided by Intravascular Ultrasound
Brief Title: Assessment of Cutting-Balloon Angioplasty With Everolimus-Eluting Stent(EES) in the Treatment of Coronary Calcified Lesion(CCL) Guided by Intravascular Ultrasonography(IVUS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry); Eulji University (Other); The Catholic University of Korea (Other); Hanil General Hospital, Korea (Unknown)
Responsible Party: Principal Investigator, Jon Suh, Jon Suh, MD/PhD, Principal investigator, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSuh
Record Dates: First submitted 2023-11-12; First posted 2023-12-20 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: Cutting balloon; Calcified coronary lesion; Calcium modification; Balloon angioplasty; Intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Intervention group : patients who received PCI with Wolverine cutting balloon to modify calcified coronary lesion; Control group : patients who received PCI with Non-compliant balloon to modify calcified coronary lesion
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Wolverine cutting balloon group (Experimental): Patients who received PCI with Wolverine cutting balloon to modify calcified coronary lesion
  Interventions: Device: Wolverine cutting balloon
- NC(Non-compliant) balloon group (Active Comparator): Patients who received PCI with Non-compliant balloon to modify calcified coronary lesion
  Interventions: Device: Non-compliant balloon

INTERVENTIONS:
Device: Wolverine cutting balloon — As an intervention method for calcified coronary lesion modification, intervention group will undergo PCI after using the Wolverine cutting balloon for calcium modification.
  Arms: Wolverine cutting balloon group
Device: Non-compliant balloon — As an intervention method for calcified coronary lesion modification, intervention group will undergo PCI after using the Non-compliant balloon for calcium modification.
  Arms: NC(Non-compliant) balloon group

SUMMARY:
The study seeks to address the clinical question of how effectively a novel cutting balloon (Wolverine™) can modify calcified lesions for stent implantation in comparison with a non-compliant (NC) balloon, particularly when used alongside a bioabsorbable polymer-coated everolimus-eluting coronary stent (Synergy™).

Most previous researches on cutting balloons focused on only severe calcifications and had limitations such as small sample sizes with retrospective designs, emphasizing on short-term imaging outcomes. This study differs by including mild to severe calcifications and evaluating long-term clinical outcomes, intraprocedural factors, and operator convenience. It aims to provide evidence that could potentially expand the indications for cutting balloon use and inform insurance coverage policies.

The objective of the study is to test the safety and efficacy of the cutting balloon in preparing calcified coronary lesions for stent insertion compared to conventional methods.

DETAILED DESCRIPTION:
1. Background

1. Which clinical question shall be answered? Heavily calcified lesions respond poorly to conventional balloon angioplasty when stents are implanted in incompletely modified lesions, resulting in incomplete and asymmetrical stent expansion. Inadequate calcium and plaque modification is related to worse clinical outcomes. In addition, incomplete modification and preparation of calcified lesions adversely affect the number of balloons, amount of contrast, procedure time, and stent delivery failure. Periprocedural factors, such as the amount of contrast medium and procedure time, are also known to be related to adverse clinical outcomes and in-hospital complication rates. Various devices, such as cutting balloons, spiral balloons, and rotational atherectomy devices, have been used to modify calcium lesions. The cutting balloon has four blades surrounding the balloon. When the balloon is inflated, the blades initiate a score into the plaque, after which the shear force applied by the balloon inflation propagates the crack and results in lumen enlargement. However, evidence related to use of the cutting balloon for various degrees of calcified lesions is limited. In addition, despite the advantages of the cutting balloon in the treatment of calcium lesions, investigations designed to focus on intraprocedural and operator-oriented endpoints, such as the number of balloons used, procedure time, and the total amount of contrast medium used, are also rare. Moreover, bioabsorbable polymer-coated coronary stents have proven to be safe and effective for the treatment of coronary artery diseases, including calcified lesions. Therefore, in this study, the investigators aim to evaluate the safety and efficacy including intraprocedural and operator-oriented outcomes of a novel cutting balloon (Wolverine™, Boston Scientific, Natick, Massachusetts(MA), USA) compared with a non-compliant (NC) balloon in the treatment of patients with various degrees of calcified lesions, including mild to heavily calcified lesions, who are treated with intravascular ultrasound (IVUS) guided bioabsorbable polymer-coated everolimus-eluting coronary stent (Synergy™, Boston Scientific Corporation, Marlborough, MA, USA) implantation.
2. To what degree has this question already been investigated elsewhere? What are the differentiators to already published studies? The Wolverine balloon (Boston Scientific Corporation) is a novel cutting balloon mounted on a semi-compliant balloon with three or four arthrotomies bonded longitudinally to its surface. Some studies on the use of cutting balloons in the treatment of coronary arteries have been previously reported, but most of them investigated moderately or severely calcified lesions compared with NC balloons. Another limitation of previous studies is that they included a small number of patients and had a retrospective design. In addition, previous studies have mainly focused on periprocedural outcomes based on imaging studies, such as acute luminal gain and cross-sectional area(CSA) using IVUS.

   In this study, the indication of a cutting balloon is not limited to severe calcified coronary artery disease but expanded to mild calcified coronary artery disease, including in-stent restenosis(ISR), to achieve optimal preconditioning for stent implantation through active calcium modification. Apart from the acute phase per-procedural gain of calcium modification, the investigators aim to investigate the long-term endpoints such as major adverse cardiac events(MACE) with aggressive calcium modification and an appropriate type of drug-eluting stent implantation. This trial is to be conducted using a bioabsorbable polymer-coated drug-eluting coronary stent. The SYNERGY stent (Boston Scientific Corporation, Marlborough, MA, USA) is a thin strut (74 μm) of platinum-chromium metal alloy that elutes everolimus from an ultrathin (4 μm) bioabsorbable polymer applied only to the abluminal surface of the stent and resolves within 4 months. After the absorption period of the polymer, only ultrathin (<70 or 80 μm) stent struts remain, and ultrathin stent struts improve clinical outcomes in the treatment of various coronary artery diseases.

   Previously, a few studies have reported the stent crossability of novel cutting balloons for treating calcium lesions. However, studies focusing on intraprocedural operator-centric factors, such as the procedure time, amount of contrast medium, and number of balloons used, are lacking. As previously reported, periprocedural and intraprocedural factors, such as the amount of contrast medium and procedure time, are also related to adverse clinical outcomes in the complex percutaneous coronary intervention(PCI) era. As (Effect of cutting balloon after rotational atherectomy in severely calcified coronary artery lesions as assessed by optical coherence tomography) reported, the low crossability of the old model cutting balloon makes the operator hesitant to choose a cutting balloon as a first-line option in the treatment of the calcified lesion. However, the crossability of the novel cutting balloon (Wolverine™) was improved and proved to have a higher delivery success rate caused by the induction of superior crossability derived from active calcium modification. In addition, owing to the development of balloon platform technologies, there have been reports on the improvement of stent and balloon crossability in the treatment of calcium lesions with novel cutting balloons compared with old cutting or scoring balloons. In our study, the investigators additionally focus on intraprocedural and operator-centric outcomes, and the total procedure time, number of balloons, and amount of contrast medium used are set as the parameters of the secondary endpoints.

   In conclusion, this study evaluates the efficacy and safety of the novel cutting balloon (Wolverine™) compared to the NC balloon in treating patients with calcified coronary lesions undergoing PCI. It aims to provide insights into the optimal type of balloons for modifying calcium lesions. Additionally, the study seeks to broaden the application of the cutting balloon, exploring its use in a range of coronary calcified lesions from mild to severe. This comparative approach extends to assessing clinical benefits, including intraprocedural and periprocedural outcomes, as well as factors like the total number of balloons used, procedure time, and contrast amount for enhanced operator convenience. Furthermore, the study intends to demonstrate the mid- to long-term clinical advantages of using cutting balloons for aggressive modification of calcified lesions, followed by the implantation of bioabsorbable polymer-coated everolimus-eluting coronary stents (Synergy™, Boston Scientific Corporation, Marlborough, MA, USA). Lastly, given the limited insurance coverage for cutting balloons in some countries, this research also aims to substantiate their use in treating mild stenosis and ISR lesions, potentially influencing broader insurance policy inclusion.
3. Can this question only be answered by a clinical investigation? Although the use of a cutting balloon in the treatment of heavy calcified lesions has been previously proven, the investigators believe that clinical studies are needed to demonstrate the effectiveness of treatment of various calcium lesions including restenosis through this study. In addition, since it is a study that requires results through imaging tests and long-term clinical observation, it is necessary to conduct clinical research. As the basis for the safety of cutting balloons has been sufficiently proven in previous clinical studies, it is considered that there are no ethical problems.
4. Why and for whom is it important to perform this study? The investigators evaluate the efficacy and safety of the novel cutting balloon (Wolverine™) in patients with calcified coronary lesions undergoing PCI and will provide rationale for which type of balloons will optimally modify the calcium lesions. In addition, the investigators attempt to expand the indications of the cutting balloon for the treatment of mild to severe coronary calcified lesions by conducting a comparative study of the NC and cutting balloons in the treatment of calcified lesions.

   The investigators aim to investigate the clinical benefits of intraprocedural and periprocedural outcomes and operator convenience, such as the number of total balloons used, procedure time, and amount of contrast. The scope of insurance coverage for cutting balloons remains limited in some countries; therefore, this study aims to provide evidence for extending insurance coverage to the treatment of mild stenosis and ISR lesions.
5. What and how will Boston Scientific technology be used? The following devices will be used: 1) Wolverine (Boston Scientific, Natick, MA, USA) cutting balloon, 2) bioabsorbable polymer-coated everolimus-eluting coronary stent (Synergy™, Boston Scientific Corporation, Marlborough, MA, USA), and 3) NC balloon (the type of NC balloon will be decided at the operator's discretion).

   PCI and stent implantation will be performed according to the current guidelines using standard interventional techniques. The interventional strategy, balloon size, and stent selection will be based on the discretion of the same operator for all patients. Modification of the atheroma using rota-ablation will be performed at the operator's discretion in cases of balloon-uncrossable lesions, and these cases will be excluded from enrollment. After pre-dilation, all patients would be treated with bioabsorbable polymer-coated everolimus-eluting coronary stent (Synergy™, Boston Scientific Corporation, Marlborough, MA, USA). After regular coronary angiography, IVUS will be performed at baseline (before pre-dilatation) and repeated immediately after stent implantation in all cases. IVUS will be performed using an OptiCross™ 60 MHz (Scientific Corporation, Maple Grove, Minnesota(MN), USA). After intracoronary injection of nitroglycerin, the IVUS catheter will be carefully advanced distal to the culprit lesion under fluoroscopic guidance and then withdrawn automatically at 0.5 mm/s to perform the imaging sequence, which begins 20 mm distal to the culprit lesion and ends at the aorto-ostial junction.
6. Is the device approved for this indication used in this study? Cutting balloon has already been approved as a treatment option for treating coronary calcified lesions. All human and animal studies were approved by the appropriate ethics committee and were, therefore, performed in accordance with the ethical standards laid down in the 1964 Declaration of Helsinki and its later amendments. In addition, this study will be approved by the ethics committee of each participating hospital and center.

2. Study Objective Calcified coronary lesions respond inappropriately to conventional balloon angioplasty, resulting in inadequate lesion preparation and incomplete stent expansion. This prospective randomized study aims to evaluate the safety and efficacy of cutting balloon angioplasty for various degrees of calcified coronary lesions treated with a novel bioabsorbable polymer-coated everolimus-eluting coronary stent.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary artery disease including ISR or de novo lesion with a stenosis of ≥ 70%
2. Target lesion calcification (an arch of calcium at least 100 degrees) was confirmed by imaging studies
3. A reference vessel diameter between 2.0 and 4.0mm and deemed suitable for PCI

Exclusion Criteria:

1. Extremely tortuous or angulated lesions
2. Lesions with dissection before balloon pre-dilatation
3. Lesions within the vein graft
4. Extremely narrow lesions which need to rotational atherectomy
5. STEMI
6. Comorbidities which preclude the achievement of one year follow up

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal stent CSA (cross-section area) with IVUS at calcium site | From date of randomization until the date of CSA(cross-section area) analysis, assessed up to one year.
  Minimal stent CSA (cross-section area) with IVUS at calcium site after modification using Wolverine cutting balloon or non-compliant(NC) balloon

SECONDARY OUTCOMES:
All-cause death | From after the index procedure up to one year.
  All-cause death during 1year follow-up after index procedure
Cardiovascular death | From after the index procedure up to one year.
  Cardiovascular death during 1year follow-up after index procedure
Myocardial infarction(MI) | From after the index procedure up to one year.
  MI during 1year follow-up after index procedure
Target vascular revascularization(TVR) | From after the index procedure up to one year.
  TVR during 1year follow-up after index procedure
Target lesion revascularization(TLR) | From after the index procedure up to one year.
  TLR during 1year follow-up after index procedure
Procedure time | From after the index procedure up to one year.
  Total procedure time of the index procedure
Total amount of contrast | From after the index procedure up to one year.
  Total amount of contrast used in the index procedure
The number of balloons | From after the index procedure up to one year.
  The total number of balloons used in the index procedure
Major adverse cardiac event(MACE) | From after the index procedure up to one year.
  MACE during 1year follow-up after index procedure
  : The number of cardiovascular death, TVR, MI will be combined to report the number of MACE

CONTACTS AND LOCATIONS:
Overall Officials: Jon Suh, PhD, Study Chair — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vavuranakis M, Toutouzas K, Stefanadis C, Chrisohou C, Markou D, Toutouzas P. Stent deployment in calcified lesions: can we overcome calcific restraint with high-pressure balloon inflations? Catheter Cardiovasc Interv. 2001 Feb;52(2):164-72. doi: 10.1002/1522-726x(200102)52:23.0.co;2-s. PMID 11170322
- [Background] Vliegenthart R, Oudkerk M, Hofman A, Oei HH, van Dijck W, van Rooij FJ, Witteman JC. Coronary calcification improves cardiovascular risk prediction in the elderly. Circulation. 2005 Jul 26;112(4):572-7. doi: 10.1161/CIRCULATIONAHA.104.488916. Epub 2005 Jul 11. PMID 16009800
- [Background] Fitzgerald PJ, Ports TA, Yock PG. Contribution of localized calcium deposits to dissection after angioplasty. An observational study using intravascular ultrasound. Circulation. 1992 Jul;86(1):64-70. doi: 10.1161/01.cir.86.1.64. PMID 1617791
- [Background] Tan K, Sulke N, Taub N, Sowton E. Clinical and lesion morphologic determinants of coronary angioplasty success and complications: current experience. J Am Coll Cardiol. 1995 Mar 15;25(4):855-65. doi: 10.1016/0735-1097(94)00462-Y. PMID 7884088
- [Background] Zaidan M, Alkhalil M, Alaswad K. Calcium Modification Therapies in Contemporary Percutaneous Coronary Intervention. Curr Cardiol Rev. 2022;18(1):e281221199533. doi: 10.2174/1573403X18666211228095457. PMID 34963434
- [Background] Aksoy A, Salazar C, Becher MU, Tiyerili V, Weber M, Jansen F, Sedaghat A, Zimmer S, Leick J, Grube E, Gonzalo N, Sinning JM, Escaned J, Nickenig G, Werner N. Intravascular Lithotripsy in Calcified Coronary Lesions: A Prospective, Observational, Multicenter Registry. Circ Cardiovasc Interv. 2019 Nov;12(11):e008154. doi: 10.1161/CIRCINTERVENTIONS.119.008154. Epub 2019 Nov 11. PMID 31707803
- [Background] Tajti P, Ayoub M, Nuehrenberg T, Ferenc M, Behnes M, Buettner HJ, Neumann FJ, Mashayekhi K. Association of Prolonged Fluoroscopy Time with Procedural Success of Percutaneous Coronary Intervention for Stable Coronary Artery Disease with and without Chronic Total Occlusion. J Clin Med. 2021 Apr 3;10(7):1486. doi: 10.3390/jcm10071486. PMID 33916666
- [Background] Feng YQ, He XY, Song FE, Chen JY. Association between Contrast Media Volume and 1-Year Clinical Outcomes in Patients Undergoing Coronary Angiography. Chin Med J (Engl). 2018 Oct 20;131(20):2424-2432. doi: 10.4103/0366-6999.243563. PMID 30334527
- [Background] Jinnouchi H, Kuramitsu S, Shinozaki T, Hiromasa T, Kobayashi Y, Takeji Y, Miura M, Masuda H, Matsumura Y, Yamaji Y, Sakakura K, Domei T, Soga Y, Hyodo M, Shirai S, Ando K. Five-Year Clinical Outcomes After Drug-Eluting Stent Implantation Following Rotational Atherectomy for Heavily Calcified Lesions. Circ J. 2018 Mar 23;82(4):983-991. doi: 10.1253/circj.CJ-17-0564. Epub 2017 Sep 9. PMID 28890526
- [Background] Li Q, He Y, Chen L, Chen M. Intensive plaque modification with rotational atherectomy and cutting balloon before drug-eluting stent implantation for patients with severely calcified coronary lesions: a pilot clinical study. BMC Cardiovasc Disord. 2016 May 26;16:112. doi: 10.1186/s12872-016-0273-8. PMID 27230875
- [Background] Karvouni E, Stankovic G, Albiero R, Takagi T, Corvaja N, Vaghetti M, Di Mario C, Colombo A. Cutting balloon angioplasty for treatment of calcified coronary lesions. Catheter Cardiovasc Interv. 2001 Dec;54(4):473-81. doi: 10.1002/ccd.1314. PMID 11747183
- [Background] Dan K, Garcia-Garcia HM, Kolm P, Windecker S, Saito S, Kandzari DE, Waksman R. Comparison of Ultrathin, Bioresorbable-Polymer Sirolimus-Eluting Stents and Thin, Durable-Polymer Everolimus-Eluting Stents in Calcified or Small Vessel Lesions. Circ Cardiovasc Interv. 2020 Sep;13(9):e009189. doi: 10.1161/CIRCINTERVENTIONS.120.009189. Epub 2020 Sep 8. PMID 32895004
- [Background] Barbato E, Shlofmitz E, Milkas A, Shlofmitz R, Azzalini L, Colombo A. State of the art: evolving concepts in the treatment of heavily calcified and undilatable coronary stenoses - from debulking to plaque modification, a 40-year-long journey. EuroIntervention. 2017 Aug 25;13(6):696-705. doi: 10.4244/EIJ-D-17-00473. PMID 28844031
- [Background] Kinoshita Y, Iwasaki K, Suzuki T. Verification of the differences of scoring effect in current scoring balloons. Cardiovasc Interv Ther. 2022 Jul;37(3):513-518. doi: 10.1007/s12928-021-00807-1. Epub 2021 Aug 25. PMID 34432207
- [Background] Zhang M, Matsumura M, Usui E, Noguchi M, Fujimura T, Fall KN, Zhang Z, Nazif TM, Parikh SA, Rabbani LE, Kirtane AJ, Collins MB, Leon MB, Moses JW, Karmpaliotis D, Ali ZA, Mintz GS, Maehara A. Intravascular Ultrasound-Derived Calcium Score to Predict Stent Expansion in Severely Calcified Lesions. Circ Cardiovasc Interv. 2021 Oct;14(10):e010296. doi: 10.1161/CIRCINTERVENTIONS.120.010296. Epub 2021 Oct 19. PMID 34665658
- [Background] Matsukawa R, Kozai T, Tokutome M, Nakashima R, Nishimura R, Matsumoto S, Katsuki M, Masuda S, Meno H. Plaque modification using a cutting balloon is more effective for stenting of heavily calcified lesion than other scoring balloons. Cardiovasc Interv Ther. 2019 Oct;34(4):325-334. doi: 10.1007/s12928-019-00578-w. Epub 2019 Feb 15. PMID 30771163
- [Background] Ishihara T, Iida O, Takahara M, Tsujimura T, Okuno S, Kurata N, Asai M, Okamoto S, Nanto K, Mano T. Improved crossability with novel cutting balloon versus scoring balloon in the treatment of calcified lesion. Cardiovasc Interv Ther. 2021 Apr;36(2):198-207. doi: 10.1007/s12928-020-00663-5. Epub 2020 Mar 28. PMID 32222901
- [Background] Tang Z, Bai J, Su SP, Wang Y, Liu MH, Bai QC, Tian JW, Xue Q, Gao L, An CX, Liu XJ. Cutting-balloon angioplasty before drug-eluting stent implantation for the treatment of severely calcified coronary lesions. J Geriatr Cardiol. 2014 Mar;11(1):44-9. doi: 10.3969/j.issn.1671-5411.2014.01.012. PMID 24748881
- [Derived] Ahn J, Yu H, Park S, Suh J. Assessment of Cutting-Balloon Angioplasty with Novel Bioabsorbable Polymer-Coated Everolimus-Eluting Stent in Treating Calcified Coronary Lesions Guided by Intravascular Ultrasound (CUPID Trial): study design and protocol. Trials. 2024 Oct 29;25(1):727. doi: 10.1186/s13063-024-08484-0. PMID 39472953

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT06177808/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT06177808/ICF_001.pdf